CLINICAL TRIAL: NCT04696640
Title: Pilot Study of Remote Glucose Monitoring Among Pediatric Patients With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 1638182
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote Patient Monitoring (Experimental): All participants who have successfully established remote data-sharing from their glucose monitors to the research team's Glooko account by conclusion of the one-month baseline period will advance to the six-month intervention period.
  Interventions: Behavioral: Remote Patient Monitoring

INTERVENTIONS:
Behavioral: Remote Patient Monitoring — Participants' glucose data will be monitored by the study team using population analytic reports. Participants who either have excessive hypoglycemia or hyperglycemia on these reports will be contacted by a pediatric endocrinologist (the principal investigator) to discuss any necessary adjustments to their home diabetes management plans. This intervention will be in addition to their usual care (regular visits at the UC Davis Pediatric Endocrinology clinic).

SUMMARY:
This project explores the feasibility and utility of remote glucose monitoring for a cohort of children and adolescents with type 1 diabetes (T1D) cared for at UC Davis Health (UCDH).

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses of type 1 diabetes with a duration of greater than or equal to 12 months
* Use of a continuous glucose monitor (CGM) for greater than or equal to 6 months
* Intention to continue receiving care at the UC Davis Health Pediatric Diabetes clinic.

Exclusion Criteria:

* Patient's CGM cannot be uploaded to Glooko

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Feasibility of remote glucose monitoring for pediatric T1D patients who receive care at UC Davis Health | 1 month baseline period
  Proportion of participants who have successfully established remote glucose monitoring by the end of the baseline period.
Change in hemoglobin A1c (HbA1c) | Initiation = 1 month after enrollment, Study completion = 7 months after enrollment
  HbA1c at study completion minus the HbA1c at initiation

SECONDARY OUTCOMES:
Data-sharing experience survey | 1 month after enrollment
  Survey asking about patient's experience with data-sharing
Target Glucose Range | Months 1-7 after enrollment
  Percentage of time spent in target glucose range (generated from continuous glucose monitor)
Hyperglycemic range | Months 1-7 after enrollment
  Percentage of time spent in hyperglycemic range (generated from continuous glucose monitor)
Hypoglycemic range | Months 1-7 after enrollment
  Percentage of time spent in hypoglycemic range (generated from continuous glucose monitor)
Overall continuous glucose monitor (CGM) wear time | Months 1-7 after enrollment
  Percentage of time spent wearing continuous glucose monitor (generated from continuous glucose monitor)
Remote patient monitoring survey | Month 7 after enrollment
  Survey asking about patient's experience with remote patient monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- University of California-Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crossen SS, Romero CC, Lewis C, Glaser NS. Remote glucose monitoring is feasible for patients and providers using a commercially available population health platform. Front Endocrinol (Lausanne). 2023 Feb 2;14:1063290. doi: 10.3389/fendo.2023.1063290. eCollection 2023. PMID 36817610
- See also: Learn more or sign up for the study here! — https://studypages.com/s/pilot-study-of-remote-glucose-monitoring-among-pediatric-patients-with-type-1-diabetes-151947/